CLINICAL TRIAL: NCT01851473
Title: Pharmacodynamic and Pharmacokinetic Interactions Between Intravenous Cocaine and Acetazolamide or Quinine
Brief Title: Interactions Between Intravenous Cocaine and Acetazolamide or Quinine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 999913482; 13-DA-N482
Record Dates: First submitted 2013-05-09; First posted 2013-05-10 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-10-07

CONDITIONS: Cocaine Use; Pharmacokinetics
Keywords: Cocaine; Pharmacokinetics; Pharmacodynamics; Drug Interactions; Acetazolamide
MeSH Terms: interventions — Cocaine; Quinine; Acetazolamide

INTERVENTIONS:
Drug: cocaine — 25 mg IV on days 1, 5, and 10
Drug: quinine — 80 mg orally on days 7-10
Drug: acetazolamide — 15 mg orally on days 2-5

SUMMARY:
Background:

- Scientists are studying medications that may be useful in treating cocaine addiction. It is important in these studies to know whether study participants are always taking their medications as directed. This study will look at two chemicals to see if they can be used to determine whether participants are taking their medications as directed. Because acetazolamide and quinine can be measured in plasma and urine, they are good test subjects for this study. They will be given alone, and combined with intravenous cocaine.

Objectives:

- To see how they body handles acetazolamide and quinine alone, and when combined with cocaine.

Eligibility:

- Individuals between 18 and 50 years of age who have smoked or used IV cocaine for at least one year and at least three times per month during the three months prior to screening. Urine test positive for cocaine within the prior 6 months

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will also be collected.
* This study will involve a 12-day inpatient stay at the National Institutes of Health.
* On days 1, 5, and 10, participants will receive a dose of cocaine. Blood, urine, breath, and saliva samples will be collected up to 18 times a day for up to about 24 hours.
* On days 2, 3, 4, and 5, participants will receive acetazolamide. Regular blood samples will be collected on Day 4.
* Day 6 is a wash-out day with no drugs or blood tests.
* On days 7, 8, 9, and 10, participants will receive quinine. Regular blood samples will be collected on Day 9.
* On day 11, blood, urine, breath, and saliva samples will be collected in the early morning. Participants will be able to leave later in the day.

DETAILED DESCRIPTION:
Background: Cocaine dependence is a public health concern worldwide, with no FDA-approved pharmacological treatment for this condition. Thus, there is a need for controlled clinical trials to evaluate potential new pharmacological treatments. Adherence to a medication regime is a major factor in the success of treatment. In controlled clinical trials, medication adherence is often monitored by measuring specific markers ingested with the medication. No such markers are validated for use in studies of cocaine dependence treatment.

Objective: Evaluate the feasibility of oral acetazolamide and quinine as adherence markers in trials of cocaine dependence treatment by determining their pharmacodynamic and pharmacokinetic interactions with intravenous (IV) cocaine.

Study Population: Up to 30 healthy cocaine users aged 18-50 years who smoked or used IV cocaine for at least one year and at least three times per month during the three months prior to screening and had a positive urine test for cocaine within the last 6 months.

Experimental Design and Methods: Participants are admitted to a secure residential research unit on and undergo baseline assessments on Day -1, receive training on Day 0, and receive single doses of IV cocaine (25 mg) on Days 1, 5 and 10. On Days 1, 5, and 10, dried blood spot specimens are collected up to 3 times daily over 1.5 h. Single oral doses of acetazolamide (15 mg) are given on Days 2-5 and quinine (80 mg) on Days 7-10. Blood, oral fluid, and breath specimens are collected for up to 71 h, 70 h, and 22 h, respectively, after drug administration on Days 1, 4, 5, 9 and 10. Participants will wear the AutoSense device on Days 1, 3, 4, 5, 8, 9 and 10 for up to 12 hours each day. All voided urine is collected throughout the study.

Outcome measures: Primary outcome measures include cocaine, benzoylecgonine, ecgonine methylester, norcocaine, acetazolamide, and quinine pharmacokinetics in plasma and urine and whether subjective and cardiovascular responses to IV cocaine are changed when coadministered with oral acetazolamide or quinine. Secondary outcome measures include cocaine pharmacokinetics in oral fluid and breath, plasma activity of BChE and carboxylesterase (enzymes which metabolize cocaine), and basal and post-cocaine administration serum concentrations of leptin and other appetitive peptides (e.g. ghrelin, GLP-1, insulin, PYY, amylin).

Benefits: There is no direct benefit to participants, but the study is likely to yield generalizable knowledge about the feasibility of acetazolamide and quinine as markers of medication adherence in future studies of pharmacological treatment for cocaine dependence.

Risks: <TAB>This study poses greater than minimal risk for participants because of IV cocaine administration.

ELIGIBILITY:
* INCLUSION CRITERIA

Age 18-50 years old

Smoked or used IV cocaine for at least six months and at least three times per month during the three months prior to screening. Urine test positive for cocaine within the prior 6 months

Adequate venous access for catheter placement

Serum sodium and potassium concentrations within normal limits (based on Johns Hopkins Bayview Medical Center clinical laboratory)

Women with reproductive potential must use a medically acceptable form of contraception for the duration of the study. Medically acceptable forms of contraception include: oral contraceptive, intrauterine device (IUD), depot hormonal preparation (ring, injection implant), or a barrier method of contraception such as a diaphragm, sponge with spermicide, or a condom.

EXCLUSION CRITERIA

Current physical dependence on any drug other than cocaine, caffeine, or nicotine

Current clinically significant medical or psychiatric disorder, such as heart disease, kidney disease, liver disease, adrenal insufficiency, myasthenia gravis, glucose-6-phosphate dehydrogenase deficiency, epilepsy, stroke, optic neuritis, hyperthyroidism, glaucoma; or psychosis, panic attacks, depression, or mania

Current sulfa allergy

Currently seeking treatment for a cocaine use disorder or in such treatment within the prior 3 months

Current hypertension or blood pressure readings consistently above 140 mm Hg systolic or 90 mmHg diastolic while at rest

Heart rate consistently above 90 bpm or below 50 bpm while at rest

History of premature coronary artery disease or heart attack before age 50 in a first degree biological relative

QTc greater than 450 ms or evidence of heart block, ischemia, or other clinically significant cardiovascular disease on a 12-lead resting ECG with three-minute rhythm strip

Hemoglobin less than 12.5 g/dL

Blood donation within 8 weeks of study entry

History of clinically significant adverse reaction to ingestion of cocaine, acetazolamide, or quinine

Hypersensitivity to acetazolamide, sulfonamides, sulfonamide derivatives, quinine, mefloquine or quinidine

Women who are pregnant or nursing

Currently on anti-hypertensive medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-10-24; Primary Completion 2015-10-07 (Actual); Study Completion 2015-10-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic changes for IV cocaine, acetazolamide, quinine | 24 hours
Heart rate, blood pressure | 3 hours
Subjective response to IV cocaine | 3 hours

SECONDARY OUTCOMES:
Esterase activity in plasma | 4 days
Pharmacokinetic parameters for IV cocain in oral fluid | 24 hours
Window of dectection for cocaine in oral fluid and exhaled breath | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Huestis, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Alboliras ET, Porter CJ, Ritter DG, Danielson GK, Driscoll DJ. Progressive atrioventricular block during exercise in univentricular heart. Pacing Clin Electrophysiol. 1986 Nov;9(6):821-5. doi: 10.1111/j.1540-8159.1986.tb06631.x. PMID 2432484
- [Background] Osterberg L, Blaschke T. Adherence to medication. N Engl J Med. 2005 Aug 4;353(5):487-97. doi: 10.1056/NEJMra050100. No abstract available. PMID 16079372
- [Background] Dubbert PM, King A, Rapp SR, Brief D, Martin JE, Lake M. Riboflavin as a tracer of medication compliance. J Behav Med. 1985 Sep;8(3):287-99. doi: 10.1007/BF00870315. PMID 4087291
- [Derived] Bouhlal S, Ellefsen KN, Sheskier MB, Singley E, Pirard S, Gorelick DA, Huestis MA, Leggio L. Acute effects of intravenous cocaine administration on serum concentrations of ghrelin, amylin, glucagon-like peptide-1, insulin, leptin and peptide YY and relationships with cardiorespiratory and subjective responses. Drug Alcohol Depend. 2017 Nov 1;180:68-75. doi: 10.1016/j.drugalcdep.2017.07.033. Epub 2017 Aug 31. PMID 28881319